CLINICAL TRIAL: NCT05484739
Title: Heat Waves in the Elderly: Reducing Thermal and Cardiovascular Consequences
Brief Title: Heat Waves and the Elderly - Cooling Modalities
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Craig Crandall, Professor of Internal Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: STU-2022-0625
Record Dates: First submitted 2022-07-27; First posted 2022-08-02 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Aging; Hyperthermia
Keywords: aging; heat wave; cardiovascular; low-energy cooling
MeSH Terms: conditions — Hyperthermia | interventions — CCP110 protein, human

STUDY DESIGN:
Intervention Model Description: The investigators will conduct a randomized crossover design study. Older individuals will be exposed to one of two heat wave conditions (Very hot and dry or hot and humid). For each heat wave condition the individual will receive one of the following cooling strategies, with each cooling strategy applied on a different day: A) a control trial, B) skin wetting only trial, C) fan only trial, and D) a combination of skin wetting with a fan trial. Thus, to complete the trial for a selected heat wave condition (e.g., either very hot and dry or hot and humid) four experimental visits will be required - one visit for each cooling strategy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Very hot and dry (Experimental): Subjects will be exposed to 3 hours in a climate chamber set to approximately 47 deg C and 15% relative humidity, which reflects a very hot and dry heat wave condition similar to the 2018 Los Angeles heat wave. Four visits will be required to complete this arm, with each visit a different cooling modality applied.
  Interventions: Other: Water Spray; Other: Fan; Other: Water Spray and Fan; Other: Control
- Hot and humid (Experimental): Subjects will be exposed to 3 hours in a climate chamber set to approximately 41 deg C and 40% relative humidity, which reflects hot and humid heat wave similar to the 1995 Chicago heat wave. Four visits will be required to complete this arm, with each visit a different cooling modality applied.
  Interventions: Other: Water Spray; Other: Fan; Other: Water Spray and Fan; Other: Control

INTERVENTIONS:
Other: Water Spray — Participants will receive water spraying on their body throughout the climate chamber exposure.
Other: Fan — Participants will be exposed to a fan throughout the climate chamber exposure.
Other: Water Spray and Fan — Participants will receive both water spraying and a fan throughout the climate chamber exposure.
Other: Control — Participants will NOT receive either water spray or a fan exposure.

SUMMARY:
The purpose of this study is to assess how well cooling modalities work in reducing cardiovascular stress of the elderly to heat wave conditions

DETAILED DESCRIPTION:
Heat waves are lethal and cause a disproportionate number of deaths in the elderly relative to any other age group. Such deaths are primarily cardiovascular, not hyperthermia itself, in origin. The central hypothesis of this work is that cardiovascular stress during heat wave conditions in the elderly can be reduced by applying low-energy cooling modalities. Comprehensive cardiovascular and thermal responses in the elderly will be evaluated during exposure to two prolonged heat wave conditions: hot and humid (replicating the 1995 Chicago heat wave), very hot and dry (replicating the 2018 Los Angeles heat wave). With each of these heat wave conditions individuals will be exposed to the following cooling modalities: no cooling (control), water spray, fan use, and fan use plus water spray.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or older
* Free of any significant underlying medical problems based upon a detailed medical history and physical exam

Exclusion Criteria:

* Known heart disease
* Other chronic medical conditions requiring regular medical therapy including cancer, diabetes, uncontrolled hypertension, and uncontrolled hypercholesterolemia etc;
* Abnormality detected on routine screening suggestive of provokable ischemia or previously undetected cardiac disease or resting left bundle branch block on screening electrocardiogram.
* Current smokers, as well as individuals who regularly smoked within the past 3 years
* Subject with a body mass index ≥31 kg/m2
* Pregnant individuals

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-02-21 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in core body temperature | Body core temperature will be obtained within 60 min before the heat wave exposure after the 3 hour heat wave exposure.
  Change in core body temperature will be measured either from a temperature sensor pill or from a rectal thermometer
Change in left ventricular function | Within 60 minutes before each simulated heat wave exposure, around minute 90 of the heat wave exposure, and at the end of the 3 hour heat wave exposure
  Measures of left ventricular function, such as ventricular wall motion and ventricular filling, will be obtained from echocardiography images.

SECONDARY OUTCOMES:
Heart rate | Prior to and throughout each simulated heat wave exposure; approximately 420 minutes
  Heart rate will be measured from ECG electrodes attached to the participant
Cardiac output | Within 60 minutes before each simulated heat wave exposure and during each simulated heat wave exposure (up to 3 hours)
  Cardiac output (how much blood is ejected from the heart) will be measured using 3D echocardiography.
Arterial blood pressure | Prior to and throughout each simulated heat wave exposure; an average of 480 minutes
  Arterial blood pressure will be measured using a standard arm blood pressure cuff.
Whole body sweat rate | Within 60 minutes before each simulated heat wave exposure and within 30 minutes after each heat wave exposure.
  Whole body sweat rate will be measured by through nude weight of the participant.
Markers of renal function and injury - Cystatin C | Within 60 minutes before each simulated heat wave exposure, during each simulated heat wave exposure (up to 3 hours), and within 2 hours after the simulated heat wave exposure
  Markers of renal function and injury (e.g., cystatin C) will be evaluated from blood sampling collection.
Markers of renal function and injury - Creatinine Clearance | Within 60 minutes before each simulated heat wave exposure, during each simulated heat wave exposure (up to 3 hours), and within 2 hours after the simulated heat wave exposure
  Markers of renal function and injury (e.g., creatinine clearance) will be evaluated from blood sampling and urine collection.
Markers of renal function and injury - Insulin-like growth factor-binding protein 7 | Within 60 minutes before each simulated heat wave exposure, during each simulated heat wave exposure (up to 3 hours), and within 2 hours after the simulated heat wave exposure
  Markers of renal function and injury (e.g., Insulin-like growth factor-binding protein 7) will be evaluated from urine sampling.
Markers of renal function and injury - Tissue inhibitor of metalloproteinases 2 | Within 60 minutes before each simulated heat wave exposure, during each simulated heat wave exposure (up to 3 hours), and within 2 hours after the simulated heat wave exposure
  Markers of renal function and injury (e.g., Tissue inhibitor of metalloproteinases 2) will be evaluated from urine sampling.
Cerebral perfusion | Within 60 minutes before each simulated heat wave exposure and during each simulated heat wave exposure (up to 3 hours)
  Cerebral perfusion will be measured by Doppler ultrasound of the internal carotid and vertebral arteries.
High sensitive cardiac troponin | Within 60 minutes before each simulated heat wave exposure, during each simulated heat wave exposure (up to 3 hours), and within 2 hours after the simulated heat wave exposure
  A plasma-based marker of cardiac stress (high sensitive cardiac troponin) be evaluated from blood sampling.
Skin temperature | Within 60 minutes before each simulated heat wave exposure and during each simulated heat wave exposure (up to 3 hours)
  Skin temperature will be measured from small temperature sensitive electrodes attached to the participant's skin
Forced vital capacity (FVC) | Within 60 minutes before each simulated heat wave exposure and during each simulated heat wave exposure (up to 3 hours)
  Forced vital capacity will be obtained from spirometry

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Health Presbyterian Hospital Dallas, Dallas, Texas, United States